CLINICAL TRIAL: NCT06568029
Title: Construct Validity and Responsiveness of EQ-5D-3L in Patients With Rheumatic Disease
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Emelie Heintz, Associate professor, Karolinska Institutet
Other Study IDs: 2023-04394-01
Record Dates: First submitted 2024-08-19; First posted 2024-08-23 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis; Polyarthritis; Psoriatic Arthritis; Ankylosing Spondylitis; Rheumatic Diseases
Keywords: EQ-5D; Validity; Responsiveness; Psychometric; Patient-reported outcome; PROM; EQ VAS
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Arthritis, Psoriatic; Spondylitis, Ankylosing; Rheumatic Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patient with rheumatoid arthritis: 18 years and older at the time of first included measurement. A diagnosis of RA. Complete registration of responses in the EQ-5D-3L descriptive system or EQ VAS on at least one time point in SRQ.
  At least one measurement with Disease Activity Score 28 (DAS28) reported in relation to the same visit as EQ-5D-3L.
  Interventions: Other: Questionnaire
- Patient with polyarthritis: 18 years and older at the time of first included measurement. A diagnosis of polyarthritis. Complete registration of responses in the EQ-5D-3L descriptive system or EQ VAS on at least one time point in SRQ.
  At least one measurement with DAS28 reported in relation to the same visit as EQ-5D-3L.
  Interventions: Other: Questionnaire
- Patients with psoriatic arthritis: 18 years and older at the time of first included measurement. A diagnosis of psoriatic arthritis. Complete registration of responses in the EQ-5D-3L descriptive system or EQ VAS on at least one time point in SRQ.
  At least one measurement with DAS28 or Disease Activity in Psoriatic Arthritis (DAPSA) reported in relation to the same visit as EQ-5D-3L.
  Interventions: Other: Questionnaire
- Patient with ankylosing spondylitis: 18 years and older at the time of first included measurement. A diagnosis of ankylosing spondylitis. Complete registration of responses in the EQ-5D-3L descriptive system or EQ VAS on at least one time point in SRQ.
  At least one measurement with the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) reported in relation to the same visit as EQ-5D-3L.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — In the study, the validity and responsiveness of EQ-5D-3L will be assessed. The EQ-5D-3L measures HRQoL and consists of two parts. The first part contains five questions about mobility, daily activities, self-care, pain/discomfort, and anxiety/depression (EuroQoL 1990, Brooks 1996). Each question can be answered with no problem (1), some/moderate problem (2) unable to perform certain activities/having extreme problems (3). The answers can be summarized in an index value based on an existing preference-based value set. In this study, the EQ-5D-3L value set by Dolan (Dolan 1997) will be used for the main analyses and a Swedish experience-based value set in a sensitivity analysis (Burström, Sun et al. 2014). For the EQ-5D-3L index, 1 represents full health and 0 represents a value equal to being dead. EQ VAS measures the persons health today on a visual analogue scale (VAS) from 0 (worst imaginable health) to 100 (best imaginable health) (EuroQoL 1990, Brooks 1996).
  Other Names: EQ-5D-3L

SUMMARY:
The aim of this study is to investigate the construct validity (convergent and known-groups) and responsiveness of EQ-5D-3L in patients with rheumatoid arthritis, polyarthritis, psoriatic arthritis, and ankylosing spondylitis. The study is based on retrospective registry data from the Swedish Rheumatology Registry (SRQ).

DETAILED DESCRIPTION:
Background

Patient-reported outcome measures (PROMs) are used to measure how patients themselves experience their health and health related quality of life (HRQoL) (Sveriges kommuner och regioner 2023). One of the most commonly used PROMs is EQ-5D, which is a generic instrument used to measure, value and compare health across symptoms and diagnoses (Devlin and Brooks 2017). When choosing a PROM to follow-up care from the patient perspective and to assess HRQoL in patients with rheumatic disease, it is important to know that the instrument is valid and responsive. An instrument with low validity and responsiveness might not capture and describe patients' health and changes in their health accurately. The aim of the study is therefore to investigate the validity and responsiveness of EQ-5D-3L. The research questions are: 1. What is the construct validity of EQ-5D-3L in patients with rheumatic disease? 2. What is the responsiveness of EQ-5D-3L in patients with rheumatic disease?

Methodology

Study design and data collection

This study will assess the construct validity and responsiveness of EQ-5D-3L among patients with rheumatoid arthritis (RA), polyarthritis, psoriatic arthritis (PsA), and ankylosing spondylitis (AS) based on retrospective registry data. The design of the study will follow the established guidelines from COSMIN on how to assess validity and responsiveness of PROMs (Mokkink, Prinsen et al. 2019).

Construct validity refers to the degree to which an instrument measures the constructs it intends to measure (Fayers and Machin 2007). Construct validity will be assessed in two ways, convergent validity and known-groups validity. Convergent validity refers to how well the instrument under study (EQ-5D-3L and EQ VAS) correlates with other outcome measures (Fayers and Machin 2007). Known-groups validity refers to how well the instrument can find differences between groups known to differ. Responsiveness refers to the ability of the instrument to capture change over time in the construct that is measured (Mokkink, Terwee et al. 2010).

Historical registry data from the Swedish Rheumatology Register (SRQ) will be used to assess the construct validity and responsiveness of EQ-5D-3L and EQ VAS. Data on EQ-5D-3L has been collected since 2008 (Ernstsson, Janssen et al. 2020) and the study will include data from 2008 until the time of data extraction. The analyses will be conducted independently for the different patient groups.

Ethical approval has been granted for the project (2023-04394-01).

Outcome measures

EQ-5D-3L and EQ VAS (see text about intervention). DAS28, DAPSA, BASDAI, ASDAS. The Health Assessment Questionnaire Disability Index (HAQ-DI), the Bath Ankylosing Spondylitis Functional Index (BASFI) VAS questions (pain, fatigue, and global score)

Convergent validity EQ-5D-3L

Convergent validity will be assessed by testing hypotheses regarding the expected direction and magnitude of correlation between the EQ-5D-3L and the other outcome measures (see hypotheses in document Study Protocol and Statistical Analysis Plan). Constructs that are considered to be related are expected to have at least a moderate correlation and constructs that are considered to be similar are expected to have a strong correlation (Prinsen, Mokkink et al. 2018).

Known-groups validity EQ-5D-3L

In the assessment of known-groups validity, patients will be divided into groups for which there is an expected difference in HRQoL (see hypotheses in document Study Protocol and Statistical Analysis Plan). The groups represent patients with different levels of disease activity or functional ability.

Responsiveness EQ-5D-3L

Responsiveness will be assessed in two ways. One way is by assessing the relationship between individual changes in EQ-5D-3L index value and dimensions over time with changes in other outcome measures over the same time period (see hypotheses in document Study Protocol and Statistical Analysis Plan). The second way is to assess whether EQ-5D-3L can discriminate between patients who have improved over time and those that have not, based on changes in disease activity or functional ability. The relationship between changes in the EQ-5D-3L and changes in other outcome measures will be assessed by analysing the correlation between the changes in the variables between the two first measurements of each individual during the first year after diagnosis (see hypotheses in document Study Protocol and Statistical Analysis Plan).

To assess whether EQ-5D-3L can discriminate between patients who have improved and those that have not, the area under the receiver operating curve ROC curve (AUC) will be calculated. Patients will be considered to have improved based on results from the measures of disease activity (DAS28, DAPSA, ASDAS or BASDAI) and functional ability (BASFI and HAQ-DI) using criteria for what is defined as a response from previous studies (see hypotheses in document Study Protocol and Statistical Analysis Plan).

Convergent validity EQ VAS

Convergent validity of EQ VAS will be assessed with the same analyses used for EQ-5D-3L (see the section about convergent validity EQ-5D-3L and hypotheses in document Study Protocol and Statistical Analysis Plan).

Known-groups validity EQ VAS

Known-groups validity of EQ VAS will be assessed for the same groups as the EQ-5D-3L index (see section about Known-groups validity EQ-5D-3L and hypotheses in document Study Protocol and Statistical Analysis Plan).

Responsiveness EQ VAS

Responsiveness of EQ VAS will be assessed with the same analyses used for EQ-5D-3L (see the section about responsiveness EQ-5D-3L and hypotheses in document Study Protocol and Statistical Analysis Plan).

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older at the time of first included measurement
* A diagnosis of RA, polyarthritis, PsA, or AS
* Complete registration of responses in the EQ-5D-3L descriptive system or EQ VAS on at least one time point in SRQ
* For patients with RA: At least one measurement with Disease Activity Score 28 (DAS28) reported in relation to the same visit as EQ-5D-3L
* For patients with polyarthritis: At least one measurement with DAS28 reported in relation to the same visit as EQ-5D-3L
* For patients with PsA: At least one measurement with DAS28 or Disease Activity in Psoriatic Arthritis (DAPSA) reported in relation to the same visit as EQ-5D-3L
* For patients with AS: At least one measurement with the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) reported in relation to the same visit as EQ-5D-3L

For the analyses of construct validity, the latest measurement will be used if the individual patients have multiple complete registrations with EQ-5D-3L and the other required measure. The hypotheses for responsiveness will be tested in patients with newly diagnosed disease (having the diagnosis for ≤12 months), as changes in disease activity are likely to be present in this group. For the analysis of responsiveness, the two first measurements during the first year will be used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is based on retrospective registry data from the Swedish Rheumatology Registry (SRQ) and includes patients with rheumatoid arthritis, polyarthritis, psoriatic arthritis, and ankylosing spondylitis. The analyses will be conducted independently for the different patient groups.
Sampling Method: Non-Probability Sample
Enrollment: 77651 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Convergent validity | One measurement per patient.The latest complete EQ-5D-3L and EQ VAS measurements per patient during the period 2008-2024 is used for the analysis.
  Convergent validity refers to how well the instrument under study (EQ-5D-3L and EQ VAS) correlates with other outcome measures (Fayers and Machin 2007). According to COSMIN guidelines, convergent validity should be assessed by formulating and testing hypotheses regarding the expected direction and magnitude of the correlation between the measurement being studied (EQ-5D-3L and EQ VAS) and other outcome measures measuring the same or similar constructs (Mokkink, Prinsen et al. 2019). The constructs measured by the other outcome measures should be clearly described (Mokkink, Prinsen et al. 2019). See hypotheses in document Study Protocol and Statistical Analysis Plan.
Known-groups validity | One measurement per patient. The latest complete EQ-5D-3L and EQ VAS measurements per patient during the period 2008-2024 is used for the analysis.
  Known-groups validity refers to how well the instrument can find differences between groups known to differ. Known-groups validity should be assessed by formulating and testing hypotheses regarding expected directions and magnitude of the differences between subgroups (Mokkink, Prinsen et al. 2019). See hypotheses in document Study Protocol and Statistical Analysis Plan.
Responsiveness | One year. The two first EQ-5D-3L and EQ VAS measurements of patients with newly diagnosed disease (having the diagnosis for ≤12 months) during the first year for patients included during the period 2008-2024
  Responsiveness refers to the ability of the instrument to capture change over time in the construct that is measured (Mokkink, Terwee et al. 2010). According to COSMIN guidelines, responsiveness can be assessed by comparing changes in EQ-5D-3L and EQ VAS, with changes in other outcome measures, similar to convergent validity explained above (Mokkink, Prinsen et al. 2019). The hypotheses should include the expected direction and magnitude of the correlations, and the constructs should be clearly described. Responsiveness can also be assessed by analysing weather EQ-5D-3L and EQ VAS can discriminate between patients who have improved and those that have not, based on changes in another outcome, such as changes in disease activity or functional ability (Mokkink, Prinsen et al. 2019). See hypotheses in document Study Protocol and Statistical Analysis Plan.

CONTACTS AND LOCATIONS:
Overall Officials: Emelie Heintz, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- It is an observational study based on the The Swedish Rheumatology Quality Register, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aletaha D, Smolen JS. The Simplified Disease Activity Index (SDAI) and Clinical Disease Activity Index (CDAI) to monitor patients in standard clinical care. Best Pract Res Clin Rheumatol. 2007 Aug;21(4):663-75. doi: 10.1016/j.berh.2007.02.004. PMID 17678828
- [Background] Boonen A, van der Heijde D, Landewe R, van Tubergen A, Mielants H, Dougados M, van der Linden S. How do the EQ-5D, SF-6D and the well-being rating scale compare in patients with ankylosing spondylitis? Ann Rheum Dis. 2007 Jun;66(6):771-7. doi: 10.1136/ard.2006.060384. Epub 2007 Jan 9. PMID 17213254
- [Background] Bruce B, Fries JF. The Stanford Health Assessment Questionnaire: dimensions and practical applications. Health Qual Life Outcomes. 2003 Jun 9;1:20. doi: 10.1186/1477-7525-1-20. PMID 12831398
- [Background] Brooks R. EuroQol: the current state of play. Health Policy. 1996 Jul;37(1):53-72. doi: 10.1016/0168-8510(96)00822-6. PMID 10158943
- [Background] Burstrom K, Sun S, Gerdtham UG, Henriksson M, Johannesson M, Levin LA, Zethraeus N. Swedish experience-based value sets for EQ-5D health states. Qual Life Res. 2014 Mar;23(2):431-42. doi: 10.1007/s11136-013-0496-4. Epub 2013 Aug 22. PMID 23975375
- [Background] Calin A, Nakache JP, Gueguen A, Zeidler H, Mielants H, Dougados M. Defining disease activity in ankylosing spondylitis: is a combination of variables (Bath Ankylosing Spondylitis Disease Activity Index) an appropriate instrument? Rheumatology (Oxford). 1999 Sep;38(9):878-82. doi: 10.1093/rheumatology/38.9.878. PMID 10515650
- [Background] Campbell, M., D. Machin and S. Walters (2007). Medical Statistics, Wiley-Blackwell.
- [Background] Coolican, H. (2014). Research methods and statistics in psychology, 6th ed. New York, NY, US, Psychology Press.
- [Background] Copay AG, Subach BR, Glassman SD, Polly DW Jr, Schuler TC. Understanding the minimum clinically important difference: a review of concepts and methods. Spine J. 2007 Sep-Oct;7(5):541-6. doi: 10.1016/j.spinee.2007.01.008. Epub 2007 Apr 2. PMID 17448732
- [Background] Devlin NJ, Brooks R. EQ-5D and the EuroQol Group: Past, Present and Future. Appl Health Econ Health Policy. 2017 Apr;15(2):127-137. doi: 10.1007/s40258-017-0310-5. PMID 28194657
- [Background] Dolan P. Modeling valuations for EuroQol health states. Med Care. 1997 Nov;35(11):1095-108. doi: 10.1097/00005650-199711000-00002. PMID 9366889
- [Background] Ernstsson O, Janssen MF, Heintz E. Collection and use of EQ-5D for follow-up, decision-making, and quality improvement in health care - the case of the Swedish National Quality Registries. J Patient Rep Outcomes. 2020 Sep 16;4(1):78. doi: 10.1186/s41687-020-00231-8. PMID 32936347
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Fayers, P. M. and D. Machin (2007). Quality of life : the assessment, analysis and interpretation of patient-reported outcomes. Chichester, J. Wiley.
- [Background] Fries JF, Spitz P, Kraines RG, Holman HR. Measurement of patient outcome in arthritis. Arthritis Rheum. 1980 Feb;23(2):137-45. doi: 10.1002/art.1780230202. PMID 7362664
- [Background] Fritz CO, Morris PE, Richler JJ. Effect size estimates: current use, calculations, and interpretation. J Exp Psychol Gen. 2012 Feb;141(1):2-18. doi: 10.1037/a0024338. Epub 2011 Aug 8. PMID 21823805
- [Background] Lukas C, Landewe R, Sieper J, Dougados M, Davis J, Braun J, van der Linden S, van der Heijde D; Assessment of SpondyloArthritis international Society. Development of an ASAS-endorsed disease activity score (ASDAS) in patients with ankylosing spondylitis. Ann Rheum Dis. 2009 Jan;68(1):18-24. doi: 10.1136/ard.2008.094870. Epub 2008 Jul 14. PMID 18625618
- [Background] Mokkink LB, de Vet HCW, Prinsen CAC, Patrick DL, Alonso J, Bouter LM, Terwee CB. COSMIN Risk of Bias checklist for systematic reviews of Patient-Reported Outcome Measures. Qual Life Res. 2018 May;27(5):1171-1179. doi: 10.1007/s11136-017-1765-4. Epub 2017 Dec 19. PMID 29260445
- [Background] Mokkink LB, Terwee CB, Patrick DL, Alonso J, Stratford PW, Knol DL, Bouter LM, de Vet HC. The COSMIN study reached international consensus on taxonomy, terminology, and definitions of measurement properties for health-related patient-reported outcomes. J Clin Epidemiol. 2010 Jul;63(7):737-45. doi: 10.1016/j.jclinepi.2010.02.006. PMID 20494804
- [Background] Nell-Duxneuner VP, Stamm TA, Machold KP, Pflugbeil S, Aletaha D, Smolen JS. Evaluation of the appropriateness of composite disease activity measures for assessment of psoriatic arthritis. Ann Rheum Dis. 2010 Mar;69(3):546-9. doi: 10.1136/ard.2009.117945. Epub 2009 Sep 17. PMID 19762363
- [Background] Prevoo ML, van 't Hof MA, Kuper HH, van Leeuwen MA, van de Putte LB, van Riel PL. Modified disease activity scores that include twenty-eight-joint counts. Development and validation in a prospective longitudinal study of patients with rheumatoid arthritis. Arthritis Rheum. 1995 Jan;38(1):44-8. doi: 10.1002/art.1780380107. PMID 7818570
- [Background] Prinsen CAC, Mokkink LB, Bouter LM, Alonso J, Patrick DL, de Vet HCW, Terwee CB. COSMIN guideline for systematic reviews of patient-reported outcome measures. Qual Life Res. 2018 May;27(5):1147-1157. doi: 10.1007/s11136-018-1798-3. Epub 2018 Feb 12. PMID 29435801
- [Background] Schoels M, Aletaha D, Funovits J, Kavanaugh A, Baker D, Smolen JS. Application of the DAREA/DAPSA score for assessment of disease activity in psoriatic arthritis. Ann Rheum Dis. 2010 Aug;69(8):1441-7. doi: 10.1136/ard.2009.122259. Epub 2010 Jun 4. PMID 20525844
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752
- [Background] Terwee CB, Prinsen CAC, Chiarotto A, Westerman MJ, Patrick DL, Alonso J, Bouter LM, de Vet HCW, Mokkink LB. COSMIN methodology for evaluating the content validity of patient-reported outcome measures: a Delphi study. Qual Life Res. 2018 May;27(5):1159-1170. doi: 10.1007/s11136-018-1829-0. Epub 2018 Mar 17. PMID 29550964
- [Background] Thyberg I, Dahlstrom O, Bjork M, Arvidsson P, Thyberg M. Potential of the HAQ score as clinical indicator suggesting comprehensive multidisciplinary assessments: the Swedish TIRA cohort 8 years after diagnosis of RA. Clin Rheumatol. 2012 May;31(5):775-83. doi: 10.1007/s10067-012-1937-0. Epub 2012 Jan 17. PMID 22249375
- See also: National Ankylosing Spondylitis Society. (2004). "Ankylosing Spondylitis (Axial Spondyloarthritis) (AS) The Bath Indices." — https://nass.co.uk/wp-content/uploads/2018/09/Bath-Indices.pdf.
- See also: Lindqvist, U. (2022). "Axial spondylartrit (ankyloserande spondylit, pelvospondylit, Bechterews sjukdom)." — https://www.internetmedicin.se/reumatologi/axial-spondylartrit-ankyloserande-spondylit-pelvospondylit-bechterews-sjukdom.
- See also: Lindqvist, U. (2022). "Psoriasisartrit." — https://www.internetmedicin.se/reumatologi/psoriasisartrit.
- See also: Mokkink, L., C. Prinsen, D. Patrick, K. Alonso, L. Bouter, H. de Vet and C. Terwee. (2019). "COSMIN Study Design checklist for Patient-reported outcome measurement instruments." — https://www.cosmin.nl/wp-content/uploads/COSMIN-study-designing-checklist_final.pdf
- See also: Svensk Reumatologis Kvalitetsregister (SRQ). "PER - Patientens Egen Registrering." — https://srq.nu/om-per-patient/
- See also: Svensk Reumatologisk Förening. (2022). "Riktlinjer för läkemedelsbehandling vid axial spondylartrit och psoriasisartrit 2022" — https://svenskreumatologi.se/wp-content/uploads/2023/01/riktlinjer-axial-spondylartrit-och-psoriasisartrit-220127.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT06568029/Prot_SAP_000.pdf